CLINICAL TRIAL: NCT02406105
Title: An Evaluation of Effectiveness and Toxicity of CyberKnife Based Functional Radiosurgery for Parkinson Disease Patients Suffering From Tremor and Its Implementation in Poland
Brief Title: An Effectiveness and Toxicity of CyberKnife Based Radiosurgery for Parkinson Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSRSPD-COI-03
Record Dates: First submitted 2015-02-22; First posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson Disease
Keywords: tremor; Parkinson disease; functional radioablation; Cyber Knife radiosurgery
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiosurgical thalamotomy (Experimental): Cyber Knife based functional radiosurgical thalamotomy, photons 6MV, single dose 70-110 Gy
  Interventions: Radiation: Radiosurgical thalamotomy; Drug: CyberKnife

INTERVENTIONS:
Radiation: Radiosurgical thalamotomy — Cybernetic microradiosurgery based thalamotomy
Drug: CyberKnife

SUMMARY:
Clinical objective of the study is estimation of effectiveness and safety of Cyber Knife based functional radiosurgery for Parkinson disease patients suffering from tremor.

DETAILED DESCRIPTION:
Basic treatment patients with Parkinson's disease (PD - Parkinson's disease) or essential tremor (ET - essential tremor) is a pharmacotherapy. In the case of lack of its effectiveness, the gold standard procedure is deep brain stimulation (DBS). Despite the proven efficacy, still remains a group of patients not eligible for this treatment. in such cases, ablation within the deep structures of the brain (thalamotomy, subthalamotomy, pallidotomy) can be considered.

Thermoablation and radiosurgery (SRS - Stereotactic radiosurgery) are used: SRS is prefered for patients who are not candidates for invasive procedures.

27 patients will be enrolled in this study. All patients will be immobilized in thermoplastic masks and planned (RT) on the base of CT/MRI fusion.

The initial total dose in the target volume (thalamic nuclei complex - VoP and VoA ) will be 70 Gy given in one fraction. The dose will be escalated every 5 Gy and the treatment effect and possible side effects will be evaluated. Dose escalation will be finished at a dose at which the effect of treatment will be satisfactory, or if side effects are unacceptable. The highest dose tested dose will be 110 Gy. Three patients will be irradiated with particular doses and observed at least 3 moths; then study will be continued.

Patients will be controlled 3, 6, 9, 12, 18 months after treatment completion and, next every each 6 months. Neurologic and neuropsychologic status, local effect (MRI ) and eventual toxicity will be checked during follow-up (FU).

ELIGIBILITY:
Inclusion Criteria:

* Idiopatic Parkinson Disease (PD)
* Lack of effective pharmacotherapy
* Lack of possibilities of qualifications to DBS (deep brain stimulation) procedure
* Informed consent for participation in the study and for radiotherapy

Exclusion Criteria:

* Age under 18
* Pregnancy
* Other than PD induced tremor
* Dementia, psychosis.
* Poor performance status
* Atrophic cerebral changes, structural changes in basal nuclei
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Tremor reduction evaluated using Unified Parkinson's Disease Rating Scale | 1 year
  Tremor reduction will be evaluated using Unified Parkinson's Disease Rating Scale (UDPRS)

SECONDARY OUTCOMES:
Safety of treatment (evaluated using RTOG/EORTC Acute Radiation Morbidity Scoring Criteria and Late Radiation Morbidity Scoring Schema) | 1 year
  Safety of treatment will be evaluated using RTOG/EORTC Acute Radiation Morbidity Scoring Criteria and Late Radiation Morbidity Scoring Schema
Evaluation of the value of magnetic resonance spectroscopy as a tool for metabolites proportions changes after PD radiosurgery (spectra of metabolites in irradiated volume) | 2 years
  None grading system of serial spectroscopy dedicated for such purpose exists. We will check spectra of metabolites in irradiated volume and proportions between them, trying to form conclusions considering necrosis/gliosis forming.
Implementation of CyberKnife radiosurgery for Parkinson disease patients not eligible for other treatment modality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Miszczyk, MD, PhD, Study Director — Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology Gliwice Branch, Gliwice, Wybrzeze AK 15, Poland

REFERENCES:
- [Background] Hooper AK, Okun MS, Foote KD, Fernandez HH, Jacobson C, Zeilman P, Romrell J, Rodriguez RL. Clinical cases where lesion therapy was chosen over deep brain stimulation. Stereotact Funct Neurosurg. 2008;86(3):147-52. doi: 10.1159/000120426. Epub 2008 Mar 12. PMID 18334856
- [Background] Niranjan A, Jawahar A, Kondziolka D, Lunsford LD. A comparison of surgical approaches for the management of tremor: radiofrequency thalamotomy, gamma knife thalamotomy and thalamic stimulation. Stereotact Funct Neurosurg. 1999;72(2-4):178-84. doi: 10.1159/000029723. PMID 10853075
- [Background] Young RF, Shumway-Cook A, Vermeulen SS, Grimm P, Blasko J, Posewitz A, Burkhart WA, Goiney RC. Gamma knife radiosurgery as a lesioning technique in movement disorder surgery. J Neurosurg. 1998 Aug;89(2):183-93. doi: 10.3171/jns.1998.89.2.0183. PMID 9688111
- [Background] Stancanello J, Romanelli P, Pantelis E, Sebastiano F, Modugno N. Atlas-based functional radiosurgery: early results. Med Phys. 2009 Feb;36(2):457-63. doi: 10.1118/1.3056460. PMID 19291984
- [Background] LEKSELL L. The stereotaxic method and radiosurgery of the brain. Acta Chir Scand. 1951 Dec 13;102(4):316-9. No abstract available. PMID 14914373
- [Background] Lindquist C, Kihlstrom L, Hellstrand E. Functional neurosurgery--a future for the gamma knife? Stereotact Funct Neurosurg. 1991;57(1-2):72-81. doi: 10.1159/000099557. PMID 1725560
- [Background] Young RF, Vermeulen S, Posewitz A, Shumway-Cook A. Pallidotomy with the gamma knife: a positive experience. Stereotact Funct Neurosurg. 1998 Oct;70 Suppl 1:218-28. doi: 10.1159/000056425. PMID 9782254
- [Background] Duma CM, Jacques DB, Kopyov OV, Mark RJ, Copcutt B, Farokhi HK. Gamma knife radiosurgery for thalamotomy in parkinsonian tremor: a five-year experience. J Neurosurg. 1998 Jun;88(6):1044-9. doi: 10.3171/jns.1998.88.6.1044. PMID 9609299
- [Background] Young RF, Jacques S, Mark R, Kopyov O, Copcutt B, Posewitz A, Li F. Gamma knife thalamotomy for treatment of tremor: long-term results. J Neurosurg. 2000 Dec;93 Suppl 3:128-35. doi: 10.3171/jns.2000.93.supplement. PMID 11143229
- [Background] Niranjan A, Kondziolka D, Baser S, Heyman R, Lunsford LD. Functional outcomes after gamma knife thalamotomy for essential tremor and MS-related tremor. Neurology. 2000 Aug 8;55(3):443-6. doi: 10.1212/wnl.55.3.443. PMID 10932286
- [Background] Okun MS, Stover NP, Subramanian T, Gearing M, Wainer BH, Holder CA, Watts RL, Juncos JL, Freeman A, Evatt ML, Schuele SU, Vitek JL, DeLong MR. Complications of gamma knife surgery for Parkinson disease. Arch Neurol. 2001 Dec;58(12):1995-2002. doi: 10.1001/archneur.58.12.1995. PMID 11735773
- [Background] Friehs GM, Park MC, Goldman MA, Zerris VA, Noren G, Sampath P. Stereotactic radiosurgery for functional disorders. Neurosurg Focus. 2007;23(6):E3. doi: 10.3171/FOC-07/12/E3. PMID 18081480
- [Background] Duma CM. Movement disorder radiosurgery--planning, physics and complication avoidance. Prog Neurol Surg. 2007;20:249-266. doi: 10.1159/000100168. PMID 17317994
- [Background] Kondziolka D, Ong JG, Lee JY, Moore RY, Flickinger JC, Lunsford LD. Gamma Knife thalamotomy for essential tremor. J Neurosurg. 2008 Jan;108(1):111-7. doi: 10.3171/JNS/2008/108/01/0111. PMID 18173319
- [Background] Young RF, Li F, Vermeulen S, Meier R. Gamma Knife thalamotomy for treatment of essential tremor: long-term results. J Neurosurg. 2010 Jun;112(6):1311-7. doi: 10.3171/2009.10.JNS09332. PMID 19895197
- [Background] Ohye C, Higuchi Y, Shibazaki T, Hashimoto T, Koyama T, Hirai T, Matsuda S, Serizawa T, Hori T, Hayashi M, Ochiai T, Samura H, Yamashiro K. Gamma knife thalamotomy for Parkinson disease and essential tremor: a prospective multicenter study. Neurosurgery. 2012 Mar;70(3):526-35; discussion 535-6. doi: 10.1227/NEU.0b013e3182350893. PMID 21904267
- [Background] Lim SY, Hodaie M, Fallis M, Poon YY, Mazzella F, Moro E. Gamma knife thalamotomy for disabling tremor: a blinded evaluation. Arch Neurol. 2010 May;67(5):584-8. doi: 10.1001/archneurol.2010.69. PMID 20457958
- [Background] Franzini A, Marchetti M, Brait L, Milanesi I, Messina G, Forapani E, Broggi G, Fariselli L. Deep brain stimulation and frameless stereotactic radiosurgery in the treatment of bilateral parkinsonian tremor: target selection and case report of two patients. Acta Neurochir (Wien). 2011 May;153(5):1069-75. doi: 10.1007/s00701-011-0962-0. Epub 2011 Feb 20. PMID 21336920
- [Background] Yu C, Main W, Taylor D, Kuduvalli G, Apuzzo ML, Adler JR Jr. An anthropomorphic phantom study of the accuracy of Cyberknife spinal radiosurgery. Neurosurgery. 2004 Nov;55(5):1138-49. doi: 10.1227/01.neu.0000141080.54647.11. PMID 15509320